CLINICAL TRIAL: NCT00298753
Title: Urinary Aquaporine 2 in Patients With Syndrome of Inappropriate ADH-secretion Caused by Treatment With Antiepileptic Medicine
Status: Withdrawn | Phase: Phase 4 | Type: Interventional
Why Stopped: no patients could be recruited
Sponsor: Regional Hospital Holstebro (Other)
Allocation: Non-Randomized | Model: Parallel | Masking: None
Other Study IDs: MED.RES.HOS.2005.04/IMT
Record Dates: First submitted 2006-03-01; First posted 2006-03-03 (Estimated); Last update posted 2015-09-15 (Estimated); Status verified 2006-09

CONDITIONS: Syndrome of Inappropriate ADH-secretion

INTERVENTIONS:
Procedure: fluid restriction for 14 days (15ml fluid per kg weight)

SUMMARY:
Patients treated with the antiepileptic drug Oxcarbazepine often develop syndrome of inappropriate secretion of antidiuretic hormone(SIADH)We want to test the hypothesis, that these patients have a higher reabsorption of water during the Aquaporine2 water channels,a higher concentration of Vasopressine (AVP), and a lower clearance of water.This situation will tend to normalize, when the patients are treated with fluid restriction

DETAILED DESCRIPTION:
The purpose of the study is to determine the amount of Aquaporine2(AQP2)in the urine in patients treated with the antiepileptic drug Oxcarbazepine before and after the administration of fluid restriction

ELIGIBILITY:
Inclusion Criteria:

Age more than 18 years, both men and women, patients with epilepsia treated with Oxcarbazepine, and a Sodium content in plasma lower than 130 mmol/liter

Exclusion Criteria:

severe diseases in the heart, lungs or liver;diabetes mellitus, other not-well treated diseases in endocrine organs, cancer; unwillingness to participate

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2005-05

CONTACTS AND LOCATIONS:
Overall Officials: Erling B Pedersen, Professor, Study Chair — Holstebro Hospital, Denmark
Locations (1):
- Department of Medicine, Holstebro Hospital, Holstebro, Jutland, Denmark